CLINICAL TRIAL: NCT01907009
Title: A Phase II Study Evaluating Intravenous Melphalan With Autologous Whole Blood Stem Cell Transplantation Over Three Cycles In Patients With Castration-Resistant Prostate Cancer (MEL-CAP)
Acronym: MEL-CAP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Early termination
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR 2012 06; 2012-000351-14 (EudraCT Number); NCT02349347 (obsolete NCT alias)
Record Dates: First submitted 2013-07-22; First posted 2013-07-24 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2020-05

CONDITIONS: Castrate Resistant Prostate Cancer
MeSH Terms: interventions — Melphalan; Lenograstim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Registration. (Experimental): MELCAP study has only one arm. All suitable patients will receive 3 cycles of melphalan and lenograstim alternately.
  Patient will start with a 3 day lenograstim (at 10mcg/kg/day) to boost up the blood cell count.
  Upon reaching sufficient blood cell count, patients will undergo a venesection and roughly a pint of blood is taken. After this patients will receive first cycle of Melphalan (60mg/m2). The following day patient will receive back the previously given whole blood. A treament break of 6 days between the cycles is given. After the break the patient will be given Lenograstim (10mcg/kg/day)for 6 days (until sufficient).
  The above regimen is repeated for cycle 2 and cycle 3 with only exception of Melphalan is given at 40mg/m2. After the cycle 3, Lenograstrim is given at 263 mcg/day for 10 days.
  Upon treatment completion, patients will be followed for 2 years. If the patients show disease progression, they will start hormone therapy.
  Interventions: Drug: Melphalan; Drug: Lenograstim

INTERVENTIONS:
Drug: Melphalan — Patients will receive Melphalan in three cycles In the first cycle they recieve 60mg/m2 and then 40mg/m2 in the next two cycles.
Drug: Lenograstim — Starting Lenograstim will be at 10mcg/kg/day and between cycles at 10mcg/kgs/day.
  After the third cycle patient will receive 263mcg/day for 10 days.

SUMMARY:
The management of (castration-resistant) prostate cancer (CRPC) is becoming increasingly complex. The use of peripheral anti-androgens with gonadorelin analogues (maximum androgen blockade) is common place. Following the failure of such an approach, several strategies may be employed. Both corticosteroids and estrogens have a role and increasingly chemotherapy is being used. The demonstration of enhanced survival using 3 weekly docetaxel has meant that this is viewed by many as the standard of care for fit patients.

Melphalan is an established alkylating drug that has demonstrated some activity in CRPC, but to date, myelosuppression has prevented adequate dosing. We have recently conducted a phase I dose escalation study using melphalan and whole blood stem cell re-infusion and it shows that median overall survival is 22 months, which is higher than the median survival rate of 19 months for Docetaxel

Data from a previous phase I study has proved the successful administration of higher doses of IV Melphalan in combination with autologous blood infusion in patients with Castration-resistant prostate cancer.

Rapid falls in circulating tumour cells were seen within 2 weeks of starting Melphalan, however slow platelet recovery meant longer periods of platelet transfusion. For this study we intend to assess the efficacy of an intensified intravenous melphalan with autologous whole blood stem cell transplantation over three treatment cycles.

39 patients will be enrolled over a 3 year period and at least 17 patients need to survive progression free at least 6-months for this study to be considered positive.

Mel-CAP is a combination chemotherapy consisting of two chemotherapy drugs:

MELPHALAN and LENOGRASTIM for 3 cycles alternately.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥18 years
2. Histological diagnosis of prostate cancer
3. Progressive Castration-resistant Prostate Cancer defined as:

   * a rising PSA; or
   * development of new sites of disease in the presence of a suppressed testosterone (<1.5 nmol/l); or
   * if testosterone >1.5 nmol/l, maximum androgen blockade failure (MAB) (MAB = GnRH analogue and peripheral anti-androgen - flutamide 250 mg 3x/day or bicalutamide 50 mg/ day or cyproterone 100mg 3x/day)
4. ECOG performance status 0-2
5. Adequate haematological reserve:

   * Unsupported Hb >9.0 g/l
   * Platelets >100x109/l
   * WBC >3x109/l
   * Neutrophils >1.5x109/l
6. Renal sufficiency:

   •Creatinine <200 µmol/l
7. Hepatic sufficiency:

   * Bilirubin <30 µmol/l
   * ALT <3xULN unless due to liver metastasis
8. Able to give written informed consent and comply with the protocol study procedures

Exclusion Criteria:

1. Patients who have suffered a previous hypersensitivity reaction to melphalan
2. Patients with known hypersensitivity to lenograstim or to any of the excipients
3. History of myeloid malignancy
4. Lenograstim should not be administered concurrently with cytotoxic chemotherapy (i.e. on the same day)
5. Previous invasive carcinoma <3 years prior to study entry
6. Cardiac condition contra-indicating large volume venesection (i.e., active angina or cardiac failure)
7. Current treatment with another investigational medicinal (chemotherapeutic) product or participation in another investigational therapeutic (chemotherapy)study, at any time during the treatment period and 30 days preceding study entry.
8. Life expectancy <12 weeks
9. Unwilling or unable to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of intensified intravenous Melphalan with autologous whole blood stem cell transplantation in patients with castration resistant prostate cancer using progression free survival. | 6 months progression free survival

SECONDARY OUTCOMES:
To determine weather early falls (two weeks)in circulating tumor cells (CTC)predict the progression free survival | 2 weeks
To assess the changes in prostate specific antigen pre and post treament | 6 months
To study progression free survival and overall survival | 6 months.
To assess the effect of this schedule in reintroduction of hormone senstivity | 6 months
To study the Quality of life. | 6 months
  QLQ-30 and PR-25 questionnaires will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shamash, MD FRCP, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- St Batholowmew's Hospital NHS, London, United Kingdom